CLINICAL TRIAL: NCT02250911
Title: Care For The Cancer Caregiver: A Meaning-Based Workshop To Help Manage Caregiver Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-208
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Caregivers
Keywords: Caregivers of patients; CCC = Care for the Cancer Caregivers; MCP-C = Meaning-Centered Psychotherapy for Cancer Caregivers; 14-208

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- This web-based CCC Workshop (Experimental): The Care for the Cancer Caregivers (CCC) workshop is composed of six webcasts. The Introductory Webcast is based upon Sessions 1 and 2 of Meaning-Centered Psychotherapy for Cancer Caregivers (MCP-C) and provides participants with an introduction to the CCC Workshop, an overview of the different meaning-centered modules (i.e., legacy, choice, creativity, and connectedness), and a discussion about identity and how caregivers' identities have or have not changed since taking on this role.
  Interventions: Other: webcasts; Behavioral: Assessments
- Waitlist Control (Active Comparator): Participants randomized to the waitlist control arm will be offered what is considered "usual care" at the ACS: the provision of the ACS Telephone Hotline number (1-800- 227-2345) and direction to the ACS website (www.cancer.org) where participants can find many resources for caregivers, including links to the ACS Caregiver ToolKit. They will complete assessments at time points that correspond with the completion of assessments in the CCC Workshop arm: after consent as soon as they are able (T1), about 2 months (± 4 weeks) after T1 (T2), and about 2-3 months after T2 (T3). Upon completion of all study assessments the waitlist control arm participants will be offered the opportunity to complete the CCC Workshop.
  Interventions: Behavioral: Assessments; Other: Usual care

INTERVENTIONS:
Other: webcasts
  Arms: This web-based CCC Workshop
Behavioral: Assessments
Other: Usual care
  Arms: Waitlist Control

SUMMARY:
The purpose of this study is to gather information on how easy it is to implement the workshop, as well as whether individuals find this workshop helpful. In this study, participants will be assigned at random to one of the two study groups. Based on the information we obtain, we hope to develop an easily accessible support service for caregivers.

ELIGIBILITY:
Inclusion Criteria:

* As per self report, a current caregiver to a patient with any site or stage of cancer
* Age 18 or over
* A score of > 4 on the Distress Thermometer (DT) and indication that this distress is related in some way to the caregiving role
* In the judgment of the investigators and/or consenting professional, able to comprehend English to complete study assessments
* Able to perform informed consent
* Enrollment is open to caregivers with their own current/past cancer histories

Exclusion Criteria:

* Significant psychiatric or cognitive disturbance sufficient, in the investigator's judgment, to preclude providing informed consent.
* As per self report, unable to access a computer with Internet or unable to use a computer with Internet provided by the study
* Participated in the development and refinement of the CCC Workshop (prospective exemption X14-006)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
feasibility of this novel approach | 2 years
  which will be measured by our ability to recruit our target sample and the proportion of participants who complete the CCC Workshop. Additional indices related to this aim (acceptability) will be gathered via both quantitative (entire sample) and qualitative (with a subset of participants randomized to received the CCC Workshop) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Applebaum, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/